CLINICAL TRIAL: NCT03460795
Title: Phase 1 Clinical Trial Using Mesenchymal Stem Cell and Regulatory T Cells as Individualized Medicine to Evaluate the Safety and Efficacy in End-stage Liver Disease
Brief Title: Safety and Efficacy Study of Co-transfering of Mesenchymal Stem Cell and Regulatory T Cells in Treating End-stage Liver Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ling Lu, Principal Investigator, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJLT005
Record Dates: First submitted 2018-02-23; First posted 2018-03-09 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conventional plus MSC and Tregs treatment (Experimental)
  Interventions: Biological: MSC and Tregs

INTERVENTIONS:
Biological: MSC and Tregs — conventional plus MSC and Tregs or placebo treatment

SUMMARY:
Cirrhosis of the liver is a common clinical chronic progressive liver disease, which is a diffuse liver lesion caused by one or more causes over a long period of time or repeatedly. Nodules, abnormal spherical areas of cells, form as dying liver cells are replaced by regenerating cells. This regeneration of cells causes the liver to become hard. The potential for stem cells to differentiate into hepatocytes cells was recently confirmed. In particular, mesenchymal stem cell (MSC) transplantation has been applicated in the clinic for treat several human diseases such as liver injury and liver fibrosis displayed good tolerance and efficiency. Besides, regulatory T cells(Tregs) had been proved as an immune regualtory T cell subsets, which could reduce immune cell activation and reduce liver injury severity. The purpose of this study is to learn whether and how MSCs and Tregs can improve the disease conditions in patients with decompensated cirrhosis.

DETAILED DESCRIPTION:
Cirrhosis of the liver is a common clinical chronic progressive liver disease, which is a diffuse liver lesion caused by one or more causes over a long period of time or repeatedly. Nodules, abnormal spherical areas of cells, form as dying liver cells are replaced by regenerating cells. This regeneration of cells causes the liver to become hard. Decompensated liver cirrhosis is mainly manifested by liver function damage and portal hypertension, with multiple system involvement. Complications such as upper gastrointestinal hemorrhage, hepatic encephalopathy, secondary infection, hypersplenism, ascites, and carcinogenesis often occur in the late stage. The potential for stem cells to differentiate into hepatocytes cells was recently confirmed. In particular, mesenchymal stem cell (MSC) and Tregs transplantation had been applicated in the clinic for treat several human diseases such as liver injury and liver fibrosis displayed good tolerance and efficiency. The purpose of this study is to learn whether and how MSCs and Tregs can improve the disease conditions in patients with decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed as decompensated liver cirrhosis.
2. Hepatitis B/C Liver Cirrhosis After Viral Treatment, HBV/HCV Viral Loads Below Detection Level over six mouths, and the liver function remained below Child-pugh A grade or MELD score >10.
3. Other causes of cirrhosis, liver function compensatory incomplete. In the past year, despite active medical treatment taken, the condition has continued to increase, at least because of cirrhosis complications such as ascites, spontaneous peritonitis, gastrointestinal bleeding, and hepatic encephalopathy in hospital over one time.
4. Need to intermittently supplement albumin and apply diuretic therapy.
5. Albumin <35 g/L, total bilirubin <170 umol/L, prothrombin activity> 30%; (Prothrombin time <20 s, moderate or lower mass ascites, spontaneous peritonitis and hepatic encephalopathy (grade II or lower), Child-pugh score> 5 points).
6. There was no history of gastrointestinal hemorrhage within the last month and population with no high-risk portal hypertension and gastrointestinal bleeding was evaluated recently.
7. Unconditional acceptance of orthotopic liver transplantation.
8. Aged from 18 to 65 years.
9. Voluntarily signed informed consent form.

Exclusion Criteria:

1. A malignant tumor with liver or other organs or a history of previous cancer.
2. Complications include gastrointestinal bleeding, spontaneous peritonitis, hepatic encephalopathy, hepatorenal syndrome, and Acute infection episodes.
3. Patients with severe heart, lung, kidney or blood system diseases and failure status.
4. Pregnant or lactating women.
5. Allergic constitution.
6. There is a history of alcohol abuse, drug abuse, and failure to effectively quit.
7. Patients did not participate in other clinical trials within 4 weeks.
8. Any condition, investigator believe that patients should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Albumin (ALB) | 24 months
  The evaluation of serum levels of ALB
Alanine aminotransferase (ALT) | 24 months
  The evaluation of serum levels of ALT
Prealbumin (PA) | 24 months
  The evaluation of serum levels of PA
Total bilirubin (TB) | 24 months
  The evaluation of serum levels of TB
Direct bilirubin (DB) | 24 months
  The evaluation of serum levels of DB
Blood urea nitrogen (BUN) | 24 months
  The evaluation of serum levels of BUN
Uric acid (UA) | 24 months
  The evaluation of serum levels of UA
Serum creatinine (Scr) | 24 months
  The evaluation of serum levels of Scr

SECONDARY OUTCOMES:
Child-Pugh | 24 months
  The evaluation of Child-Pugh score for liver function
Model for end-stage liver disease (MELD) | 24 months
  The evaluation of MELD score for severity of liver disease
Quality of life (QOL) | 24 months
  The evaluation of QOL score for life quality

OTHER OUTCOMES:
Evaluation of liver fibrosis | 24 months
  The pathology decrease in grade of liver fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Tang, M.D, PH.D, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Medical University, Nanjing, Jiangsu, China